CLINICAL TRIAL: NCT04374084
Title: Moxibustion Plus Cupping in Convalescent Patients With COVID-19: A Randomized Clinical Trial
Brief Title: Moxibustion Plus Cupping in Convalescent Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Hubei Provincial Hospital of Integrated Chinese & Western Medicine (Unknown); Wuhan Hospital of Traditional Chinese Medicine (Other); Wuhan Third Hospital (Other); Huangshi Hospital of Traditional Chinese Medicine (Unknown); Yichang Hospital of Traditional Chinese Medicine (Other); Ezhou Hospital of Traditional Chinese Medicine (Unknown); Hunan University of Traditional Chinese Medicine (Other); The Hospital of Jiangxi University of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Xiaopin Wang, Secretary of Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020YFC0845000
Record Dates: First submitted 2020-04-20; First posted 2020-05-05 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Convalescence
Keywords: Moxibustion; COVID-19; Randomized Clinical Trial
MeSH Terms: conditions — COVID-19; Convalescence | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moxibustion plus Cupping (Experimental): Moxibustion plus cupping and basic therapy (rehabilitation direction and basic breathing exercise) once a day for 4 weeks (28 sessions).The moxibustion plus cupping treatments were divided into 2 alternating formulas:
  A: Monday, Wednesday, Friday and Sunday: moxibustion on bilateral Fengmen (BL12), Feishu (BL13) and Pishu(BL20) B: Tuesday, Thursday and Saturday: moxibustion on Zhongwan (RN12), Qihai (RN6), bilateral Tianshu(ST25) and Zusanli(ST36) + cupping on bilateral Feishu(BL13) Geshu(BL17) Pishu(BL20) The 2 formulas were used alternatively every other day, 7 times per week, for 4 weeks. Moxibustion acupoint addition: profuse sweating added Fuliu (KI7), insomnia added Shenmen(HT7) anxiety or depression added Neiguan (PC6).
  Interventions: Other: Moxibustion plus Cupping
- Basic therapy (No Intervention): Basic therapy: rehabilitation direction and basic breathing exercise.

INTERVENTIONS:
Other: Moxibustion plus Cupping — Moxibustion: The burning of a small, thimble sized, smoldering plug of dried leaves on the skin at an acupuncture point. Usually the plugs contain leaves of mugwort or moxa. Cupping takes the pot as a tool, uses the combustion to remove the air in the pot, causes a negative pressure, and makes it adsorb on the skin of the acupoints. Use"Baixiaojiu"moxibustion on each acupoint for 10-15 minutes, the temperature of moxibustion should be adjusted within patient's tolerance level. Use diameter of 5-6 cm acuum cupper to cupping on each acupoint for 5-8 minutes.
  Arms: Moxibustion plus Cupping

SUMMARY:
This trial is designed to evaluate the efficacy and safety of moxibustion plus cupping in the convalescence of COVID-19.

DETAILED DESCRIPTION:
Moxibustion plus cupping may be effective and safe for convalescent patients with COVID-19, but evidence is limited. The randomized clinical trial may help to provide evidence-based factors for improving the patients' symptoms in the convalescence of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of the convalescence of COVID-19 (defined by the Chinese Guideline for COVID-19 in 2020 Trial Version 7).
2. 18-70 years old;
3. chest tightness/fatigue/shortness of breath/cough, with at least 2 of the above symptoms and the average VAS score (last 48 hours) ≥ 40 points;
4. Volunteers with informed consent;

Exclusion Criteria:

1. Surgery in the lung that affects lung function;
2. Rely on mechanical ventilation to maintain lung function;
3. Chronic lung diseases affecting lung function;
4. Diseases affecting heart function;
5. Severe basic diseases;
6. Resting heart rate > 120/min, systolic blood pressure > 180mmHg, diastolic blood pressure > 100mmHg;
7. Unstable angina or myocardial infarction in the past 1 month;
8. Severe obesity (BMI>30kg/m2);
9. Allergic constitution;
10. Pregnant or lactating women;
11. Disabled patients;
12. Mentally ill Patients;
13. Participating in other clinical trials;
14. Poor compliance or other complicate conditions according to the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of responder at week 4 | baseline, week 4
  The responder is defined as the participants with ≥ 50% average VAS decrease of chest tightness and fatigue compared with baseline. The VAS ranges from 0 to 100.

SECONDARY OUTCOMES:
The proportion of responder at week 8 | baseline, week 8
  The responder is defined as the participants with ≥ 50% average VAS decrease of chest tightness and fatigue compared with baseline. The VAS ranges from 0 to 100.
The change in the average VAS score of main symptoms from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the change in the average VAS score of main clinical symptoms (chest tightness, fatigue, short of breath and cough) will be assessed from baseline. VAS ranges from 0-100.
The change in the severity VAS score of main symptoms from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the change in the severity VAS score of main clinical symptoms (chest tightness, fatigue, short of breath and cough) will be assessed from baseline. VAS score ranges from 0-100.
The change in the average VAS score of other symptoms from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the change in the average VAS score of other symptoms (insomnia, sweating, mental fatigue, inappetence, mental stress) will be assessed from baseline. VAS score ranges from 0-100.
The change in mean frequency of diarrhea and spontaneous bowel movements from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the change in mean frequency of diarrhea and spontaneous bowel movements in the past 1 week will be assessed from baseline.
The proportion of participants with ≥50%/75% improvement of VAS from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the proportion of participants with ≥50%/75% VAS change of clinical symptoms (chest tightness, fatigue, short of breath, cough, insomnia, sweating, mental fatigue, inappetence, mental stress) will be assessed. VAS score ranges from 0-100.
The change of the walking distance of six-minute-walking test from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the walking distance of six-minute-walking test changed from baseline.
The change of the lowest oxygen saturation of six-minute-walking test from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the lowest oxygen saturation of six-minute-walking test changed from baseline.
The proportion of patients in recovery of pulmonary function at week 4 | baseline, week 4
  At the end of week 4, the proportion of patients in recovery of pulmonary function in all participants.
The proportion of patients whose lung CT return to normal at week 4 | baseline, week 4
  Lung CT shows complete absorption of inflammation.
The change of the WHO QOL-BREF score from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the WHO Quality of Life-BREF (WHO QOL-BREF) score changed from baseline. WHO QOL-BREF ranged from 4 to 20 with higher scores as the better quality of life.
The change of the SAS score from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the Self-Rating Anxiety Scale (SAS) score changed from baseline. The standard SAS ranged from 25 to 100 with higher score as the worse anxiety.
The change of the SDS score from baseline | baseline, week 4, week 8
  At the end of week 4 and week 8, the Self-Rating Depression Scale (SDS) score changed from baseline.The standard SAS ranged from 25 to 100 with higher score as the worse depression.
The change of the blood CRP/LYMPH#/NEUT% value from baseline | baseline, week 4
  At the end of week 4, the blood C-reactive protein (CRP) value, blood lymphocyte count (LYMPH#) and the percentage of blood neutrophils (NEUT%) value will be assessed compared with baseline.
subtype analysis | baseline, week 4
  Subtype analysis of age (≤40 years old, >40 years old), gender (male, female), and severity of the disease (mild, moderate, heavy, critical) will be performed in the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaopin Wang, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences; Zhongyu Zhou, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (1):
- Hubei Province Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available on reasonable request. You can send e-mail to us if you have any question.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: It depends.
Access Criteria: It depends.